CLINICAL TRIAL: NCT00299351
Title: A Multicenter, Open-Label Continuation Trial Evaluating the Tolerability and Activity of Depsipeptide (FK228) in Patients That Have Completed a Prior Clinical Study With Depsipeptide.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR2742
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2006-03-06 (Estimated); Status verified 2005-11

CONDITIONS: Peripheral T Cell Lymphoma (PTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Depsipeptides

INTERVENTIONS:
Drug: Depsipeptide

SUMMARY:
To evaluate the safety and tolerability of extended treatment with depsipeptide in patients who have at least demonstrated stable disease on prior Gloucester-sponsored depsipeptide clinical trials, and in the opinion of their physician/ investigator might benefit from continued treatment with depsipeptide

ELIGIBILITY:
Inclusion Criteria:

Written informed consent/ authorization Patient has completed 6 cycles of therapy in a prior Gloucester-sponsored depsipeptide clinical trial Patient has immediate past participation (not to exceed 21 days from Day 15 of cycle 6 in the previous study) in a prior Gloucester-sponsored depsipeptide clinical trial Patient has demonstrated stable disease, partial response or complete response as best overall response in their prior Gloucester-sponsored depsipeptide clinical trial and such response must be ongoing at the time of enrollment Patient must have serum potassium levels >4.0mEq/L and serum magnesium levels >2.0mg/dL Negative urine or serum pregnancy test on females of childbearing potential Sexually active females of child-bearing potential must be willing to practice reliable methods of birth control to prevent pregnancy after entering the trial Sexually active males must be willing to practice reliable methods of birht control after entering the trial

Exclusion Criteria:

Patients wiht known cardiac abnormalities such as

* congenital long QT syndrome
* QTc interval >480 milliseconds Patients with any cardiac arrhythmia requiring anti-arrhythmic medication Patients who have had a history of coronary artery disease (CAD) eg. angina Canadian class II-IV (see appendix G)> In any patient whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiopathy to define whether or not CAD is present Patients who have had a myocardial infarction within 12 months of study entry. Patients with an ECG recorded at screening showing evidence of cardiac ishemia (ST depression of >2mm). If in any doubt, the patient should have a stress imaging study and if abnormal, angiograpphy to define whether or not CAD is present Patients with congestive heart failure that meets New York heart Association (NYHA) Class II to IV (see appendix F) definitions and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or magnetic resonance imaging (MRI) Patients with a history of sustained VT,VF,Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD) Patients with a hypertrophic cardiomelagy or restrictive cardiomyopathy from prior treatment or other causes (in doubt, see ejection fraction criteria above) Patients with uncontrolled hypertension ie > 160/95 Concomitant use of medications which may cause a prolongation of QT/QTc Concomitant use of medications that are inhibitors of the cytochrome P-450 isoenzyme CYP 3A4 Absolute neutrophil count (ANC) < 1.5 X 109 cells/L Platelet count <75 x 109 cells/L Serum creatinine concentration >2 mg/dL or creatinine clearance <40mL/min AST (aspartate aminotransferase ) and alanine aminotransferase (ALT) >2.0 x ULN or >5 X ULN in presence of demonstable liver metastasis Bilirubin concentration > 1.25 x ULN or > 2.0 x ULN in presence of demonstrable liver metastases Serum potassium <4.0mEq/L and serum magnesium <2.0 mg/dL Failure to recover of any drug-related non-hematological toxicity to grade 1 oe less or to baseline values unless otherwise indicated Concomitant use of warfarin (due to a potentialdrug to drug interaction with depsipeptide) Patient is pregnant or nursing Patient had been on prior Gloucester-sponsored depsipeptide clinical trial, left the trial and then received alternative neoplastic therapy

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8

CONTACTS AND LOCATIONS:
Overall Officials: Dr Johann De Bono, Principal Investigator — Royal Marsden NHS Foundation Trust